CLINICAL TRIAL: NCT06026046
Title: Feasibility of an Adapted Sports Program Based on Fencing to Reduce Physical Deconditioning in Adult Hematology Patients Receiving Intensive Treatment
Brief Title: Feasibility of an Adapted Sports Program Based on Fencing to Reduce Physical Deconditioning in Adult Hematology Patients
Acronym: EscrimHEMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC23_0088; 2023-A01596-39 (Other: ANSM)
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients benefiting from the adapted sport program based on fencing (Experimental)
  Interventions: Other: Adapted sport program based on fencing

INTERVENTIONS:
Other: Adapted sport program based on fencing — This adapted sport program includes 3 to 5 sessions per week of adapted fencing (excluding weekends and public holidays), carried out either by a fencing master trained in adapted sport, or by an APA teacher trained in adapted fencing by the fencing master.
  Sessions can last from 10 to 30 minutes. The course of the session is validated by the fencing master and adapted to each patient. The limiting factors are taken into account, in order to direct towards a specific practice.
  The sessions are progressive with very short and varied sequences calling on the imagination and experience of the fencing masters.

SUMMARY:
In 20 years, the prognosis of hematology patients has improved thanks to the development and adaptation of treatments and better risk management. However, medium and long-term complications of intensive treatments are common and remain a real public health problem. Indeed, intensive treatments associated with room confinement within a protected unit expose patients to physical deconditioning of multifactorial pathophysiological mechanisms. If this deconditioning is neglected, response to treatment, tolerance, quality of life and, in the longer term, survival will be impacted.

Several teams have demonstrated the feasibility and the benefits of physical support for patients with prolonged aplasia. These studies focused on peripheral stem cell allograft, which occur late in the treatment of acute leukemia. On the other hand, studies evaluating the benefits of physical support as soon as the diagnosis of acute leukemia is made and intensive treatments are started are rare. Implementing a adapted sport program from the diagnostic and throughout the course of treatment is therefore a worthwhile subject for research.

The adapted sport chosen was fencing because it responds to hematological problems. Fencing is adaptable without carrying or receiving blow, can be practiced standing up, in an armchair or in bed, involves praxis and concentration, and involves the whole body. It can be practiced individually or as part of a team, in a protected room or in a unit corridor. Fencing is a fighting sport and includes a psychological aspect, with a possible projection of a fight against the disease. In addition, fencing is carried out by a non-medical or paramedical practitioner, which can reinforce or recreate an image of normal activity. Finally, the attention required by listening to the fencing master and the necessary concentration unconsciously pushes the patient to "get out of his illness".

The aim of this pilot study is to assess the feasibility, throughout the care pathway, of an adapted sport program based on fencing in adult patients with hematological malignancies receiving intensive treatment, to reduce physical deconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to a protected unit of the Hematology department of one of the participating centers
* Patient with acute leukemia treated in induction with "3+7" or "5+7" intensive treatment or by an equivalent treatment (Vyxeos, azacitidine+vénetoclax), or patient admitted for an allograft or CAR-T cells and not included at the diagnosis of the disease
* Patient eligible for intensive chemotherapy
* Patient requiring prolonged hospitalization with room confinement
* Signed informed consent form

Exclusion Criteria:

* Patient with a neurological or cardiac disease that contraindicates the practice of fencing
* No intensive treatment with prolonged hospitalization
* Pregnant, parturient or breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person under legal protection
* Person unable to express consent
* Person not covered by or not benefiting from a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-06-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients attending at least 50% of the schedulded lessons over the entire duration of the program | 1 year
  The proportion of patients attending at least 50% of the scheduled fencing lessons over the entire duration of the program will be used to evaluate the feasibility of the adapted sport program based on fencing.

SECONDARY OUTCOMES:
Number of actual fencing lessons compared to number of scheduled fencing lessons | 1 year
  The comparison between the number of fencing lessons patients actually attended and the number of fencing lessons theoretically planned will be used to assess adherence to the adapted sport program.
Average duration of fencing lessons | 1 year
  The average duration of the program corresponds to the average duration of the adapted sport program for each participant in real-life conditions. It will be used to assess the adequacy of the theoretical modalities and the implementation of the program in real-life conditions .
Average duration of the program | 1 year
  The average duration of the program corresponds to the average duration of the adapted sport program for each participant in real-life conditions. It will be used to assess the adequacy of the theoretical modalities and the implementation of the program in real-life conditions .
Typology of patients attending at least 50% of the scheduled fencing lessons over the entire duration of the program | 1 year
  The typology of patients will be described according to pathology, age, co-morbidities, type of intensive chemotherapy, treatment phase (induction, consolidation, allograft, CAR-T cells)
Comparison between the EORTC-QLQC30 score obtained at inclusion and the score obtained at each prolonged hospitalization discharge and at 3 months, 6 months and 1 | 1 year
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer - C30 is used to assess the quality of life.
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer - C30 comprises 30 items. The 28 first items are constructed on a Likert scale with 4 response modalities (1 "Not at all" / 2 "A little" / 3 "Quite a lot" / 4 "A lot"), the modality 4 representing a high level of symptomatology / problems. The last two items are constructed on a 7-modality scale. These two items respectively assess overall health and overall quality of life, with response modality 1 corresponding to a "very poor" state, and response modality 7 to an "excellent" state.
Evolution of the distance covered in 6-minute walk test between inclusion and 6-month follow-up | 6 months
  The 6-minute walk test is used to assess functional exercise capacity of an individual. It measures the distance an individual is able to walk over a 6-minute period.
Evolution of the SPPB (Short Physical Performance Battery) score between inclusion and 6-month follow-up | 6 months
  The SPPB test is used to assess the physical performance of an individual. Il is the result of the scores of three criteria: the balance test, the walking speed test and the sit-to-stand test. The sum of the scores of all the tests gives an overall performance score.
Evolution of the upper limb grip strength measured by dynamometer between inclusion and 6-month follow-up | 6 months
  This test is used to measure muscle strength in the hand and forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Aline MD Schmidt, PHD, Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - University Hospital, Angers, Angers
  - University Brest Hopspital, Brest

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).